CLINICAL TRIAL: NCT00594464
Title: An Explorative, Multicenter, Open-label Pilot Trial With Neupro® (Rotigotine Transdermal Patch) Once Daily Treatment Administered Perioperatively in Patients With Idiopathic Parkinson's Disease
Brief Title: A Trial of Neupro® (Rotigotine Transdermal Patch) in Patients With Parkinson's Disease Undergoing Surgery
Acronym: NEUPOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0882; 2006-005438-19 (EudraCT Number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-15 (Estimated); Results first posted 2009-07-03 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2010-12

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine; NEUPRO®; Parkinson's Disease (PD); perioperative use; anaesthesia,
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Rotigotine
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — 2 mg/24 h, 4 mg/24 h, 6 mg/24 h and 8 mg/24 h patch;
  Single patches and a combination of 2 of these patches for a dosage of up to 16 mg/24 h;
  One (1) regimen on day of surgery, but exceptionally extended for up to 2 (two) weeks if the patient requires unexpected ventilation after surgery.

SUMMARY:
Evaluation of efficacy and safety on the use of rotigotine in patients suffering from Parkinson's Disease during and after surgery requiring general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has idiopathic Parkinson's disease (early- or advanced-stage), as defined by the cardinal sign bradykinesia, plus the presence of at least one of the following: resting tremor, rigidity, or postural instability and is without any other known or suspected cause of Parkinsonism.
* Subject is scheduled for an operation requiring general anesthesia.

Exclusion Criteria:

* Subject has previously been treated with rotigotine.
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermals or recent unresolved contact dermatitis or has a known allergy or hypersensitivity to rotigotine or to other components of the patch.
* Subject is scheduled for a surgical procedure (surgery per protocol(SPP)) that requires magnetic resonance imaging or cardioversion.
* Subject has a high probability to require extended postoperative ventilation (> 24 hours).
* Subject has any medical condition that, in the opinion of the investigator, could jeopardize or compromise the subject's ability to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (12):
- Germany (12):
  - Augsburg
  - Bochum
  - Bonn
  - Bremerhaven
  - Dortmund
  - Dresden
  - Hanau
  - Ingolstadt
  - Kiel
  - Schwerin
  - Stralsund
  - Ulm

REFERENCES:
- [Result] Wullner U, Kassubek J, Odin P, Schwarz M, Naumann M, Hack HJ, Boroojerdi B, Reichmann H; NEUPOS Study Group. Transdermal rotigotine for the perioperative management of Parkinson's disease. J Neural Transm (Vienna). 2010 Jul;117(7):855-9. doi: 10.1007/s00702-010-0425-4. Epub 2010 Jun 10. PMID 20535621
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotigotine: Patients were dispensed rotigotine patches up to 16mg/24h at a dose left to the discretion of the neurologist.
Period: Overall Study
Arm/Group | Rotigotine
Started | 14
Completed | 11
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Delay in operation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  Germany | 14

OUTCOME MEASURES:

1. Primary Outcome: Efficacy and Safety of Rotigotine Used During Surgery Under General Anaesthesia Assessed by Anaesthesiologist.
Description: Questionnaire including 4 items Range of sum score: 4 to 24 Range of item scores: 1 (I agree completely) to 6 (I don't agree at all) Item 1: Patient did not show unexpected symptoms Item 2: Handling was simple Item 3: Handling wasn't time-consuming Item 4: Patch is a considerable option
Time Frame: After subject wakes up from general anesthesia
Population: Full Analysis Set (Subjects having valid data for all three feasibility assessments)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 9
Score on scale | 5.0 (1.8)

2. Secondary Outcome: Plasma Concentration of Rotigotine After Use.
Time Frame: 24 hours
Population: Pharmacokinetic Set (Subjects for whom a blood sample for determination of the plasma concentration of rotigotine was drawn and a valid determination of the plasma concentration could be done)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Rotigotine 2 mg/24h | Rotigotine 6mg/24h | Rotigotine 8 mg/24h | Rotigotine 12 mg/24h | Rotigotine 14 mg/24h | Rotigotine 16 mg/24h
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 1 | 3
ng/ml | 0.1640 (0) | 0.2480 (0) | 0.7570 (0.1569) | 0.8405 (0.3302) | 0.8689 (0) | 1.6958 (2.1951)

3. Primary Outcome: Efficacy and Safety of Rotigotine Used During Surgery Under General Anaesthesia Assessed by Neurologist.
Description: Questionnaire including 4 items Range of sum score: 4 to 24 Range of item scores: 1 (I agree completely) to 6 (I don't agree at all) Item 1: Switch to patch was easily feasible Item 2: Re-switch was easily feasible Item 3: Patient did not show unexpected symptoms Item 4: Patch is a feasible option
Time Frame: 2 weeks after surgery
Population: Full Analysis Set (Subjects having valid data for all three feasibility assessments)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 9
Score on scale | 5.2 (2.2)

4. Primary Outcome: Efficacy and Safety of Rotigotine Used During Surgery Under General Anaesthesia Assessed by Patient.
Description: Questionnaire including 3 items Range of sum score: 3 to 18 Range of item scores: 1 (I agree completely) to 6 (I don't agree at all) Item 1: Therapy with patch was easily feasible Item 2: Symptoms of Parkinson's Disease were well controlled Item 3: I felt safe with the Parkinson patch
Time Frame: 2 weeks after surgery
Population: Full Analysis Set (Subjects having valid data for all three feasibility assessments)
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 9
Score on scale | 3.9 (1.4)

ADVERSE EVENTS:
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=14)
Ventricular asystole (Cardiac disorders) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4)
Staphylococcal infection (Infections and infestations) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
Urine uric acid increased (Investigations) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (3)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.